CLINICAL TRIAL: NCT06730321
Title: Surgical Competency for Robot-Assisted Thyroidectomy: Construction and Validation of a Robotic Thyroidectomy Assessment Score (RTAS)
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Doctor, Shanghai 6th People's Hospital
Other Study IDs: 2024-KY-245(K)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Cancer; Thyroid Nodule; Thyroid Diseases; Thyroid Cancer, Papillary; Thyroid Cancer, Follicular
Keywords: Robotic thyroidectomy; Surgical competency; Robotic thyroidectomy assessment score
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Thyroid Diseases; Thyroid Cancer, Papillary; Thyroid cancer, follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent robotic thyroidectomy: Patients underwent robotic thyroidectomy without conversion during the study period
  Interventions: Other: Observations on clinicopathological factors influencing the assessment score of surgery

INTERVENTIONS:
Other: Observations on clinicopathological factors influencing the assessment score of surgery — Age, body mass index, gender, thyroid function parameters, lesion size, lesion location, ultrasound data

SUMMARY:
To develop and validate a structured scoring tool (robotic thyroidectomy assessment score, RTAS) for assessing and quantifying surgical performance in robotic thyroidectomy (RT).

DETAILED DESCRIPTION:
This study was conducted in two phases. In the first phase, the content development and validation phase, the key elements of robotic thyroidectomy with central neck dissection were broken down into 9 key steps for assessing the technical skills required to complete the procedure: creating the surgical area, exposing the thyroid gland, dissecting the upper pole of the thyroid gland with preservation of the superior laryngeal nerve (SLN), identifying and protecting the upper pole of the parathyroid glands, protecting the retractor laryngeal nerve (RLN), identifying and protecting the lower pole of the parathyroid glands, removing the thyroid, dissection of the central neck region and hemostasis.

The Delphi method was used for content validation of the 9 key steps. Each item was described using a Likert scale: 1 for worst and 5 for best. Experts were invited to evaluate each of the 9 key steps in terms of the description of the items and the agreement of the items with the assigned scores. Based on the Delphi method, the opinions of the experts were collected and consensus on the entry was indicated by determining that a content validity index (CVI) > 0.75 (CVI measure: the proportion of experts who scored each entry 4 or 5. Consensus is considered to have been reached when the CVI reaches 0.75. For entries where consensus was not reached entries were revised to reflect any changes suggested by the expert group and the revised scoring system was recirculated for reassessment. This process is repeated until all entries have reached consensus.

In the second phase of the study, the structural validation phase, two consecutive 50 robotic by the same operator after a learning curve were scored. The aim was to analyze whether the scoring system developed in the first phase could assess operator progress and steps for improvement. In addition, the time taken to complete the procedure was recorded and compared. It was also analyzed whether there were any differences in the baseline (tumor size, location, age, gender, etc.) of the patients in the two groups (1st 50 cases and 2nd 50 cases).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of differentiated thyroid cancer with a maximum diameter not exceeding 4 cm
* Clinical diagnosis of benign thyroid nodules with a maximum diameter not exceeding 6 cm
* Participants with high cosmetic expectations
* Participants underwent robotic thyroidectomy without open conversion

Exclusion Criteria:

* Participants with history of neck surgery or radiation
* Participants with vocal fold fixation by preoperative fibrolaryngoscope
* Participants with preoperative examination suggestive of distant invasion
* Participants with fusion or fixed of lymph nodes in the neck

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were well informed about the robotic thyroidectomy and were aware of the potential benefits and risks. Patients underwent robotic thyroidectomy during the study period. Patient consented for us to use perioperative data.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with recurrent laryngeal nerve injury | through study completion, an average of 1 year
  impaired vocal cord mobility confirmed by postoperative laryngoscopy
Number of participants with hypoparathyroidism | through study completion, an average of 1 year
  a postoperative parathyroid hormone level of less than 10 pg/ml
Operative time | through study completion, an average of 1 year
  operative time was defined as the duration from incision to closure, and was collected from anesthesia record sheet
Score for surgical competence | at the end of robotic thyroidectomy
  score evaluated by the proposed assessment system

SECONDARY OUTCOMES:
hospitalization | through study completion, an average of 1 year
  days of hospitalization
degree of pain | approximately 4 hours after surgery and on postoperative day 1
  pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, Doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided